CLINICAL TRIAL: NCT02442037
Title: Safety and Efficacy of Human Umbilical-Cord-derived Mesenchymal Stem Cell Transplantation in Active Ulcerative Colitis.
Brief Title: Human Umbilical-Cord-Derived Mesenchymal Stem Cell Therapy in Active Ulcerative Colitis
Acronym: UCMSC-UC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Collaborators: Ivy Institute of Stem Cells Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 307-IVY-SC-002
Record Dates: First submitted 2015-05-06; First posted 2015-05-13 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Ulcerative Colitis
Keywords: cellular therapy; active ulcerative colitis; phase 1/2 clinical study; human umbilical cord mesenchymal stem cell; allogeneic stem cell transplantation; UC
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UCMSC group (Experimental): Human umbilical cord MSCs are administrated to patients by three intravenous infusion
  Interventions: Biological: UCMSC group
- Control group(Normal saline) (Other): Patients will receive normal saline at the same time points as that in experimental group.
  Interventions: Other: Control group(Normal saline)

INTERVENTIONS:
Biological: UCMSC group — Human umbilical cord MSCs are transplanted three times by intravenous infusion(1×10^6/kg) ,once every week，a total of three times.
  Arms: UCMSC group
Other: Control group(Normal saline) — Normal saline in same volume as MSCs are transplanted to patients.
  Arms: Control group(Normal saline)

SUMMARY:
Phase I-II Clinical Trial - Safety and efficacy of umbilical-cord-derived mesenchymal stem cell (UC-MSC) in patients with active ulcerative colitis，randomized, single blind, controlled prospective study.

DETAILED DESCRIPTION:
Phase I-II Clinical Trial - Safety and efficacy of umbilical-cord-derived mesenchymal stem cell (UC-MSC) in patients with active ulcerative colitis，randomized, single blind, controlled prospective study.

Thirty patients will be selected and randomized into two groups: the first group of 15 patients will receive a sole injection of UC-MSC and the remaining 15 patients will comprise the control group.

Every patient will maintain their standard treatment of active ulcerative colitis, with maximum tolerated dosage without side effects.

The day of infusion will be considered day zero. From that moment, followup will be divided into 0-1 week, 1 week-2 week,2 week-3 week, 3 week-1 month, and 3 month-6 months.

Clinical results will be analyzed after completion of 6 months of followup.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of active UC must have been confirmed by endoscopic and histological evidence.
* With mild and moderate disease.
* Men and women 18-65 years of age.
* Signed informed consent
* Capable of good communication with researchers and follow the entire test requirements

Exclusion Criteria:

* Patient with associated diseases such as diabetes mellitus, hypertension, dyslipidemia, atherosclerosis and malabsorption syndrome.
* With autoimmune diseases (lupus, HIV, cancer and hepatitis), colitis (infectious, post-radiation, post-drug, indeterminate) and Crohn's Disease.
* Abnormal hepatic or renal function
* Prior history of malignancy
* Pregnant or unwilling to practice contraceptive therapy or breast feeding females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety will be determined by the assessment of major adverse events. | Within the six months after intravenous infusion
  Safety will be determined by the assessment of major adverse events defined as fever, allergy or any other intravenous infusion adverse events.

SECONDARY OUTCOMES:
Clinical response (CDAI points) | Post first cell transplantation: 3 weeks and months 1,3 and 6
  CDAI is defined as Clinical Disease Activity Index.
Endoscopic improvement is assessed by UCEIS. | Post first cell transplantation 6 months
  UCEIS is defined as Ulcerative Colitis Endoscopic Index of Severity.
Level of C-reactive protein | Post first cell transplantation: 3 weeks and months 1,3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Bing Liu, M.D., Study Chair — 307-IVY Translational Medicine Center; Yan Liu, M.D., Study Director — Department of gastroenterology,Affiliated Hospital to Academy of Military Medical Sciences; Min Min, M.D., Principal Investigator — Department of gastroenterology,Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Department of gastroenterology,Affiliated Hospital to Academy of Military Medical Sciences, Beijing, China